CLINICAL TRIAL: NCT02429700
Title: A Multicenter, Prospective, Randomized Trial Comparing Paclitaxel and Carboplatin or Bleomycin, Etoposide and Cisplatin in the Treatment of Ovarian Malignant Sex Cord-Stromal Tumors
Brief Title: TC or BEP in Treating Patients With Ovarian Malignant Sex Cord-Stromal Tumors
Acronym: SCST-01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beihua Kong (Other)
Collaborators: Huazhong University of Science and Technology (Other); Zhejiang University (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, Beihua Kong, MD. PhD., Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCST-01
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Ovarian Sex Cord Stromal Tumor; Ovarian Neoplasms; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Taxes; Carboplatin; Bleomycin; Etoposide; etoposide phosphate; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PT (Arm 1) (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 1 hour on day 1. Treatment repeats every 21 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin
- BEP (Arm 2) (Active Comparator): Patients receive bleomycin IM daily for days 1-3, etoposide IV daily for days 1-5, cisplatin IV for days 1-5. Treatment repeats every 21 days for 3 or 4* courses in the absence of disease progression or unacceptable toxicity.
  NOTE: *Patients who have good risk will have 3 courses and those who have poor risks will have 4 courses.
  Interventions: Drug: Bleomycin; Drug: Etoposide; Drug: Cisplatin

INTERVENTIONS:
Drug: Paclitaxel — Patients receive paclitaxel 175mg/㎡ IV over 3 hours on day 1. Treatment repeats every 21 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: Anzatax; TAX
  Arms: PT (Arm 1)
Drug: Carboplatin — and carboplatin AUC 5-6 IV over 1 hour on day 1. Treatment repeats every 21 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.
  Arms: PT (Arm 1)
Drug: Bleomycin — Bleomycin 30000IU IM per day for 3 days every 3 weeks for 3-4 cycles.
  Other Names: Blanoxan; BLEO; BLM
  Arms: BEP (Arm 2)
Drug: Etoposide — Etoposide 100mg/㎡ IV per day for 5 days every 3 weeks for 3-4 cycles.
  Other Names: ETOP; Etopophos
  Arms: BEP (Arm 2)
Drug: Cisplatin — Cisplatin 20mg/㎡ IV per day for 5 days every 3 weeks for 3-4 cycles in the absence of disease progression or unacceptable toxicity.
  Arms: BEP (Arm 2)

SUMMARY:
Investigators will conduct the trial to determine whether paclitaxel and cisplatin (PT) has the same curative effects and less adverse effects than bleomycin, etoposide and cisplatin(BEP) among newly diagnosed ovarian malignant sex cord-stromal tumor patients after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To assess the activity of paclitaxel and carboplatin with respect to progression free survival (using bleomycin, etoposide, and cisplatin [BEP] as a reference) for newly diagnosed ovarian malignant sex cord-stromal tumors.

SECONDARY OBJECTIVES:

1. To estimate the toxicity of paclitaxel and carboplatin, and bleomycin, etoposide, and cisplatin in this patient population.
2. To estimate overall survival for paclitaxel and carboplatin relative to that of BEP.
3. To evaluate response rate in the subset of patients with measurable disease.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

ARM 1: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 1 hour on day 1. Treatment repeats every 21 days for 4-6 courses in the absence of disease progression or unacceptable toxicity.

ARM 2: Patients receive bleomycin IM daily for days 1-3, etoposide IV daily for days 1-5, cisplatin IV for days 1-5. Treatment repeats every 21 days for 3 or 4* courses in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients who have good risk will have 3 courses and those who have poor risks will have 4 courses.

Patients undergo blood sample collection at baseline and periodically during study for laboratory biomarker analysis.

After completion of study therapy, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age≤65 years; female, Chinese women;
* Histologically confirmed ovarian stromal tumor, including the following cell types:

  * Granulosa cell tumor
  * Granulosa cell-theca cell tumor
  * Sertoli-Leydig cell tumor (androblastoma)
  * Steroid (lipid) cell tumor
  * Gynandroblastoma
  * Unclassified sex cord-stromal tumor
  * Sex cord tumor with annular tubules
* Newly diagnosed, stage IIA-IVB disease;

  * Has undergone initial surgery (for diagnosis, staging, or cytoreduction) within the past 8 weeks.
  * May or may not have measurable residual disease.
* Laboratory tests: WBC≥4×10(9)/L, NEU≥2×10(9)/L, PLT≥80×10(9)/L, serum bilirubin≤ 1.5 times the upper limit of normal, transaminase≤ 1.5 times the upper limit of normal, BUN, Cr≤ normal
* Performance status: Karnofsky score≥60;
* Provide written informed consent.

Exclusion Criteria:

* With severe or uncontrolled internal disease, unable to receive surgery and/or unsuitable for chemotherapy;
* History of organ transplantation, immune diseases;
* History of serious mental illness, a history of brain dysfunction;
* Drug abuse or a history of drug abuse;
* Suffering from other malignancies;
* Concurrently participating in other clinical trials
* Unable or unwilling to sign informed consents;
* Unable or unwilling to abide by protocol.

Ages: 14 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2015-04; Primary Completion 2025-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Date of randomization, and death due to any cause, assessed up to 5 years
  PFS was definite as the time from randomization to disease recurrence (including death from recurrence if it was the first manifestation of recurrence), death without recurrence.

SECONDARY OUTCOMES:
Chemotherapy related adverse effects in two arms | Up to 5 years
Tumor response rate | Up to 5 years
  The relationship of treatment to tumor response rate will be assessed using logistic regression models adjusted for age and stratification factor (measurable disease status).
Overall survival | Up to 5 years
  The relationship of treatment to overall survival will be assessed using the proportional hazards model.

CONTACTS AND LOCATIONS:
Overall Officials: Beihua Kong, MD. PhD., Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China